CLINICAL TRIAL: NCT07098481
Title: Access to Hepatitis C Treatment in Cameroon: Comparison of a Simplified Test and Treat Strategy to a Standard Strategy
Acronym: ACCESS+
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: IRD, Epidemiologie et Prevention, Montpelier, France (Unknown); SESSTIM (IRD, Inserm, Université Aix-Marseille) (Unknown); Centre de Recherche sur les Maladies Emergentes et Re-Emergentes (CREMER) (Unknown); Faculté de Médecine et des Sciences Biomédicales, Université de Yaoundé I, Yaoundé, Cameroun (Unknown); PharmAccess (Unknown); Service d'hépato-gastroentérologie, Hôpital Saint Joseph, Marseille, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 0388s ACCESS+
Record Dates: First submitted 2025-07-01; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hepatitis C Virus Infection
Keywords: simplified test and treat strategy; hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: two-arm, cluster-randomized, controlled phase 4 trial will be conducted in blood banks and HIV clinics (the clusters) in the two largest cities in Cameroon (Yaoundé and Douala).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACCESS+ Strategy (Experimental): ACCESS+ strategy will rely on four components:
  1. same-day on-site rapid anti-HCV and HCV RNA testing,
  2. same-day on-site pan-genotypic DAA treatment initiation,
  3. minimal clinical and biological monitoring, and
  4. management by trained general medical doctors and counselors (community health workers, nurses or social workers) in non-specialist services.
  Interventions: Drug: ACCESS+ strategy Epclusa 400/100 Oral Tablet; Drug: ACCESS+ Strategy Vosevi 400/100/100 Oral Tablet
- Standard Strategy (Experimental): In the standard strategy based on routine medical practice in Cameroon, anti-HCV positive participants will be referred to and managed by gastroenterologists, and the patients' management will be closer. However, the process for screening and treatment initiation will be longer.
  Interventions: Drug: Standard Strategy Vosevi 400/100/100 Oral Tablet; Drug: Standard Strategy Epclusa 400/100 Oral Tablet

INTERVENTIONS:
Drug: ACCESS+ strategy Epclusa 400/100 Oral Tablet — The ACCESS+ strategy will rely on four components: (1) same-day on-site rapid anti-HCV and HCV RNA testing (rapid diagnostic test and GeneXpert), (2) same-day on-site pan-genotypic DAA treatment initiation (sofosbuvir 400 mg/velpatasvir 100 mg once daily for 12 weeks), (3) minimal clinical and biological monitoring, and (4) management of patients in non-specialist services by trained general medical doctors and counselors (community health workers, nurses or social workers).
  Arms: ACCESS+ Strategy
Drug: ACCESS+ Strategy Vosevi 400/100/100 Oral Tablet — The ACCESS+ strategy will rely on four components: (1) same-day on-site rapid anti-HCV and HCV RNA testing (rapid diagnostic test and GeneXpert), (2) same-day on-site pan-genotypic DAA treatment initiation (sofosbuvir 400 mg/velpatasvir 100 mg/voxilaprevir 100mg) once daily for 12 weeks, (3) minimal clinical and biological monitoring, and (4) management of patients in non-specialist services by trained general medical doctors and counselors (community health workers, nurses or social workers).
  Arms: ACCESS+ Strategy
Drug: Standard Strategy Vosevi 400/100/100 Oral Tablet — In the standard strategy based on routine medical practice in Cameroon, anti-HCV positive participants will be referred to and managed by gastroenterologists who will initiate pan-genotypic DAA treatment initiation (sofosbuvir 400 mg/velpatasvir 100 mg/voxilaprevir 100mg) once daily for 12 weeks, and the patients' management will be closer. However, the process for screening and treatment initiation will be longer.
  Arms: Standard Strategy
Drug: Standard Strategy Epclusa 400/100 Oral Tablet — In the standard strategy based on routine medical practice in Cameroon, anti-HCV positive participants will be referred to and managed by gastroenterologists who will initiate pan-genotypic DAA treatment initiation (sofosbuvir 400 mg/velpatasvir 100 mg) once daily for 12 weeks, and the patients' management will be closer. However, the process for screening and treatment initiation will be longer.
  Arms: Standard Strategy

SUMMARY:
Hepatitis C is a common and potentially serious disease. However, there are treatments that can cure it. That's why it's so important to detect the hepatitis C virus (HCV) and treat those affected. Today, many hepatitis C sufferers in Cameroon (and elsewhere) remain untreated.

The aim of this research is therefore to evaluate a simplified screening and treatment strategy (developed specifically for the Cameroonian context) in comparison with a standard strategy (based on usual care), in order to improve access to hepatitis C treatment in Cameroon. If the results of this research are positive, this strategy could be recommended to health authorities in Cameroon and other comparable countries.

DETAILED DESCRIPTION:
A two-arm, cluster-randomized, controlled trial will be conducted in blood banks and HIV clinics (the clusters) in the two largest cities in Cameroon (Yaoundé and Douala).

Persons aged 21 years or older, anti-HCV positive, and living in the study area will be eligible. The ACCESS+ strategy will rely on four components: (1) same-day on-site rapid anti-HCV and HCV RNA testing, (2) same-day on-site pan-genotypic DAA treatment initiation, (3) minimal clinical and biological monitoring, and (4) management by trained general medical doctors and counselors (community health workers, nurses or social workers) in non-specialist services. In contrast, in the standard strategy, the process for screening and treatment initiation will take longer, and anti-HCV positive participants will be managed by gastroenterologists and will have a closer follow-up.

Biological and clinical data (using standardized case report forms), socioeconomic data (using standardized questionnaires), and qualitative data (using interviews and focus groups) will be collected. A total of 576 anti-HCV positive participants (288 per arm) will be recruited in 16 facilities (8 blood banks and 8 HIV clinics) after testing approximately 32,000 blood donors and 8,400 patients living with HIV. The total duration of the trial will be 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Persons of both genders aged 21 years or older
* Anti-HCV positive;
* Living in the study area
* Agreeing to participate in the trial and signing the informed consent form.

Exclusion Criteria:

* Participationin a previous study on HCV treatment
* Previous sofosbuvir treatment
* HBsAg positive or indeterminate;
* Pregnancy test positive ;
* Life-threatening condition ;
* Impairment of the person making it difficult, if not impossible, for them to participate in the trial or to understand the information given to them.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of ACCESS+ strategy | 12 weeks after the end of treatment
  % of anti-HCV positive patients at enrolment who were correctly managed (classified as follows): Success if either one of the following statement is reached 'baseline HCV RNA negative and informed of this result' or 'baseline HCV RNA positive, treated and HCV RNA negative 24 weeks after start of treatment' Failure in the other situations including 'baseline HCV RNA not tested', 'baseline HCV RNA negative but not informed of this result', 'baseline HCV RNA positive and untreated', 'baseline HCV RNA positive, treated and HCV RNA positive or not tested 24 weeks after start of treatment', and 'missing data'

SECONDARY OUTCOMES:
HCV cascade (HCV RNA Test) of care between both strategies | 12 weeks after end of treatment
  % of anti-HCV positive patients who had an HCV RNA test
HCV Cascade (HCV RNA positive) of care between both strategies | 12 weeks after end of treatment
  % of anti-HCV positive patients who were HCV RNA positive
HCV Cascade (communication of HCV RNA Status) of care between the two strategies | 12 weeks after end of treatment
  % of anti-HCV positive patients who were aware of HCV RNA status
HCV Cascade (start of treatment) of care between the two strategies | 12 weeks after end of treatment
  % of HCV RNA positive patients who started direct-acting antiviral (DAA) treatment
HCV Cascade (treatment completed) of care between the two strategies | 12 weeks after the end of treatment
  % of HCV RNA positive patients who completed the treatment; % of HCV RNA positive patients who were cured
HCV Cascade (patients cured) of care between the two strategies | 12 weeks after the end of treatment
  % of HCV RNA positive patients who were cured
Patient-reported outcomes between both strategies | 12 weeks after end of treatment
  Barriers to HCV testing and treatment reported by patients and healthcare workers through qualitative interviews
Patient-reported outcomes (quality of life) between both strategies | 12 weeks after end of treatment
  Changes in health-related quality of life in Short Form-12 scale (SF-12), giving a physical and mental health summary of the participant
Patient-reported outcomes (fatigue) between both strategies | 12 weeks after end of treatment
  Changes in fatigue reported in Fatigue scale (scale graduated from 0 to 10, with 0 corresponding to no fatigue and 10 an extreme fatigue)
Cost-effectiveness of the ACCESS+ strategy | 12 weeks after end of treatment
  Total cost of the two strategies over the trial period and over the long term, in terms of disability adjusted life years, and quality-adjusted life years

IPD SHARING:
Plan to Share IPD: Undecided